CLINICAL TRIAL: NCT01533649
Title: Pilot Trial: Personalizing Health Outcome in Epilepsy Now - An Introduction to Clinical Services
Brief Title: Personalizing Health Outcome in Epilepsy Now - An Introduction to Clinical Services
Acronym: PHOENICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHOENICS-01
Record Dates: First submitted 2012-02-06; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Medically Intractable Epilepsy
Keywords: Behavioral intervention; Seizure self-efficacy; Psychosocial outcomes; Quality of Life in Epilepsy
MeSH Terms: interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A/R intervention (Experimental): The A/R intervention will accommodate 10 study subjects who will participate in an epilepsy-specific counseling intervention.
  Interventions: Behavioral: Andrews/Reiter approach to epilepsy
- Relaxation (Experimental): The relaxation group will accommodate 10 study subjects who will participate in a condition unspecific supportive relaxation intervention.
  Interventions: Behavioral: Relaxation/Meditation
- Usual care (No Intervention): 10 Potential study subjects who are not interested in participating in either intervention will be asked to provide data as a usual care control group.

INTERVENTIONS:
Behavioral: Andrews/Reiter approach to epilepsy — The Andrews/Reiter approach to epilepsy is a systematic semi-directive, multi-modal counseling intervention that integrates conventional therapies, educational modules, psychological interventions and relaxation techniques in order to assist the individual in improving self-defined life quality. Face-to-face counseling sessions and supervision with telephone calls are based on a standardized workbook ("Taking Control of Your Epilepsy") as an on-going step-by-step guideline.
  Other Names: A/R intervention
  Arms: A/R intervention
Behavioral: Relaxation/Meditation — Subjects who participate in the relaxation control group will attend weekly relaxation sessions that will employ the following relaxation techniques: meditation, progressive muscle relaxation, autogenic training.
  Arms: Relaxation

SUMMARY:
The assumption of the unpredictability of seizures may have an enormous impact on the perception of self-efficacy and may contribute more to a patient's poor quality-of-life than the actual seizures. Patients with epilepsy are especially susceptible to the influence of the arbitrary nature of this condition on socialization,education,and the formation of self-identity. Consequentially, the psychosocial and psychological aftermath is likely to be observed even in individuals with well-controlled seizures. The relationship between seizure occurrence and the effects of having epileptic seizures on quality of life can be characterized as reciprocal; e.g. emotional stress is not only a result of having seizures; it is also the most frequently reported seizure precipitant. Whereas behavioral interventions have repeatedly been considered as the third pillar of the treatment of epilepsy, the main focus still remains on passive seizure control per pharmacological and surgical interventions, which may further aggravate victimization. Outcome after epilepsy surgery is closely correlated with pre-surgical characteristics. Consequentially, there is an upsurge of interest in the medical community for research on non-pharmacologic interventions to facilitate the transition from chronically sick to well with preventive therapeutic interventions in the context of habitual seizures. The Andrews/Reiter (AR) approach to epilepsy is a systematic counseling intervention that assists the individual to identify seizure warning signs,seizure precipitants and general life stressors in order to develop strategies of active seizure control and improve self-defined life quality. Literature review indicates that AR represents the most comprehensively developed psychological approach. The proposed trial will address the question if AR decreases seizure frequency and psychopathologic comorbidities and increases seizure self-efficacy and overall quality of life in patients with medically intractable epilepsy.

DETAILED DESCRIPTION:
Potential subjects will be systematically approached during a 3 years enrollment period to recruit a consecutive sample of the patient population receiving care at a tertiary care epilepsy center (Toronto Western Hospital). After an 8 week period to establish baseline measurements the proposed trial will allocate study subjects to an A/R intervention group or a relaxation/meditation control group or a usual care control group (N1=N2=N3=10) per their preference due to the fact that internalization of the therapeutic principles is an active process that requires continuous motivation and compliance of the patient with the intervention. If a subject displays high intrinsic motivation to engage in self-care enhancing activities but does not indicate a preference, he or she will get randomized to either the A/R intervention or the relaxation protocol. This trial design allows for measuring effect sizes in regard the potential effect of choice, and also whether there is any interaction between preference and treatment.

This trial will determine the following:

I. The fraction of (a) seizure-free subjects and (b) subjects with clinically meaningful, i.e. ≥ 90% or ≥ 50 reduction of seizure frequency, II. Changes of the subjective perception of disability as indicated by Subjective Handicap of Epilepsy Scale (SHE), III. Changes of seizure self-efficacy as indicated by Multidimensional Health Locus of Control (M-HLOC), Form C and Epilepsy Self-Efficacy Scale (ESES), IV. Changes in common psychopathologic comorbidities and stress as indicated by (a) Neurological Disorders Depression Inventory in Epilepsy (NDDI-E), (b) State Trait Anxiety Inventory (STAI), (c) Profile of Mood States (POMS brief), and (d) Perceived Stress Scale (PSS), V. Changes in quality of life as indicated by (a) Quality of Life in Epilepsy (QOLIE-89), (b) individually identified descriptors of various domains of life and (c) individually identified epilepsy-related distresses. Continuous measures (aims I and III b) will be obtained during months 9 and 10 after initial subject enrollment. All other measures will be obtained at the end of month 10.

Intervention Protocols: During months 3-5 the A/R intervention protocol devotes one face-to-face counseling session to each of the 11 chapters ("steps") of the workbook "Taking control of your epilepsy" which will be followed by weekly phone calls during months 6-8. A/R treatment plans include daily activities: Journaling (10 min), CD-guided relaxation (10-30 min), Workbook (10 min) to promote functional analysis of seizure context and development of coping strategies. The trial will be used for knowledge-translation as trainees delivering the intervention will be supervised by Donna Andrews, PhD, co-developer of the AR intervention. The relaxation and meditation protocol will consist of weekly 30 min session during months 3-5 and bi-weekly 60 min sessions during months 6-8.

All subjects are instructed to document seizure occurrences (number and type) and compliance with AEDs. They will continue to see their treating neurologist and adjustment of their antiepileptic medication will be made if necessary. Medication changes will be included in outcome analyses. Regular serum levels will be drawn to monitor drug compliance. Study subjects will be approached at 12, 24 and 36 months after the end of the pilot trial to obtain follow-up data. The sample size determination the investigators based on literature review, assuming the remission rate for the usual care group was 5% and 35% for the A/R intervention group and inflated by 30% to account for loss to non-compliance. Outcomes will be compared as found in groups as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years old
* Fluency in English, including reading and writing
* Confirmed diagnosis of epilepsy as indicated by review of medical records (video-EEG, routine EEG and imaging)
* Drug-refractoriness as indicated by at least two failures to achieve seizure freedom per adequate drug trials in the patient's history
* Eligibility to be subjected to a surgical intervention aiming at seizure reduction
* A baseline seizure frequency of at least two complex partial seizures per month
* Willingness not to begin another non-pharmaceutical treatment while enrolled in the study
* Readiness to attempt not to change pharmaceutical treatment while enrolled in the study
* Motivation to comply with the intervention protocols

Exclusion Criteria:

* A history of a relapsing remission course of epilepsy
* Presumed psychogenic events
* Scheduled or likely change of treatment within 8 months after enrollment in the trial
* Negative compliance history
* Noncompliance with baseline measurement
* A seizure frequency of less than two seizures per month during baseline measurement
* Serious other medical problems, such cancer, stroke, significant heart disease, psychiatric disorders
* Brain tumors, vascular malformations, progressive epilepsy syndromes, neurodegenerative disorders or significant developmental delay (IQ<80)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Fraction of seizure free study subjects | Change from baseline seizure frequency obtained during months 1 and 2 at months 9 and 10 after initial subject enrollment.
  The determination of the fraction of seizure-free study subjects will be the primary outcome measure of this pilot trial. Seizure freedom will be defined as absence of seizures (not auras) during months 9 and 10 after initial subject enrollment.

SECONDARY OUTCOMES:
Fraction of subjects achieving a clinically meaningful reduction of seizure frequency | Change from baseline seizure frequency obtained during months 1 and 2 at months 9 and 10 after initial subject enrollment.
  The fraction of subjects achieving a clinically meaningful reduction of seizure frequency will be determined. Reduction of seizure frequency will be categorized as ≥ 90% reduction of seizures or ≥ 50% reduction of seizures
Subjective Handicap of Epilepsy | Change from baseline questionnaire scores obtained during month 1 at month 10 after initial subject enrollment
  Changes as indicated by the completion of the subjective Handicap of Epilepsy 32-item (SHE) scale at baseline and at the end of month 10 after subject enrollment.
Health-related self-efficacy | Change from baseline questionnaire scores and fraction of days with reported side effects obtained during months 1 and 2 at months 9 and 10 after initial subject enrollment.
  Changes as indicated by the completion of the 18-item Multidimensional Health Locus of Control (M-HLOC) Questionnaire.Different aspects of efficacy in the self-management of epilepsy will be measured using the 2000 version 33-item Epilepsy Self-Efficacy Scale (ESES). The fraction of days with reported medication side effects will be determined comparing documentations obtained during the initial 8 weeks of baseline measurement with adverse event documentation obtained during months 9 and 10 after initial subject enrollment.
Psychopathologic disorders and stress | Change from baseline questionnaire scores obtained during month 1 at month 10 after initial subject enrollment.
  Changes in the 6-item Neurological Disorders Depression Inventory in Epilepsy (NDDI-E), the State Trait Anxiety Inventory (STAI), the 30-item Profile of Mood States (POMS-Brief), and the 14-item Perceived Stress Scale (PSS)
Quality of life | Change from baseline questionnaire scores obtained during month 1 at month 10 after initial subject enrollment
  Changes in regard to 89-item Quality of Life in Epilepsy (OLIE-89) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Taufik A Valiante, MD PhD FRCS, Principal Investigator — Toronto Western Hospital; University Health Networks
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Reiter JM, Andrews DJ. A neurobehavioral approach for treatment of complex partial epilepsy: efficacy. Seizure. 2000 Apr;9(3):198-203. doi: 10.1053/seiz.1999.0374. PMID 10775516
- See also: Link to Andrews/Reiter epilepsy research.inc who have been applying the studied intervention for more than 30yrs. — http://www.andrewsreiter.com/